CLINICAL TRIAL: NCT00967642
Title: Intravenous Insulin for 24 Hours in Patients With Diabetes Mellitus Submitted to Percutaneous Coronary Intervention With Stent: Effects Upon Oxidative Stress and Inflammatory Markers
Brief Title: Intravenous Insulin in Patients With Diabetes After Percutaneous Coronary Intervention (PCI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); FIPE (Unknown)
Responsible Party: Marco Vugman Wainstein/MD, HOSPITAL DE CLINICAS DE PORTO ALEGRE
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06036
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes Mellitus; Percutaneous Coronary Intervention
Keywords: Patients with Diabetes Mellitus Submitted to Percutaneous Coronary Intervention with Stent
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard treatment (No Intervention): glycemia before meals and subcutaneous regular insulin if higher than 200 mg/dl
- Intravenous Insulin (Other): intravenous insulin/24h guided by glycemia (Optium, Abbott) evaluated hourly, targeting values lower than 110 mg/dl
  Interventions: Drug: Intravenous Insulin

INTERVENTIONS:
Drug: Intravenous Insulin — continuous intravenous insulin/24h guided by glycemia (Optium, Abbott) evaluated hourly, targeting values lower than 110 mg/dl
  Arms: Intravenous Insulin

SUMMARY:
The purpose of this study is to evaluate the effects of intravenous insulin/24 hours to normalize glycemia upon markers of oxidative stress (protein oxidation and total antioxidant defense) and inflammation (C-reactive protein (CRP) and sCD40L) in diabetic patients submitted to PCI with stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetes Mellitus submitted to Percutaneous Coronary Intervention with Stent bare metal
* Age: 18-80 years old

Exclusion Criteria:

* Restenosis
* Drug elution stent
* Acute coronary syndrome at last 30 days
* Use anti inflammatory, antibiotic, vitamin E
* Inflammatory disease or oncologic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Reintervention, Myocardial Infarction, Cardiovascular Death | 6 months